CLINICAL TRIAL: NCT00737932
Title: A Phase IIa, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Sequential Cohorts, Dose Range Finding Study to Evaluate the Safety, Tolerability and Clinical Effect of Escalating Doses of Laquinimod in Active Moderate to Severe Crohn's Disease.
Brief Title: Laquinimod Phase IIa Study in Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CD-LAQ-201
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — laquinimod

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Laquinimod (Experimental): Laquinimod 0.5mg/day, 1mg/day, 1.5mg/day, 2mg/day (sequential cohorts)
  Interventions: Drug: Laquinimod
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Laquinimod — Laquinimod 0.5mg/day, 1mg/day, 1.5mg/day, 2mg/day, oral, for 8 weeks of treatment
  Arms: Laquinimod
Other: placebo — Matching placebo for 8 weeks of treatment
  Arms: Placebo

SUMMARY:
The study aims to evaluate the safety and clinical effect of daily oral treatment of Laquinimod capsules in active moderate to severe Crohn's disease. This study will assess Laquinimod doses of 0.5mg /day to 2 mg/day in sequential dose groups (cohorts). Laquinimod is a novel immunomodulating drug which is currently in advanced stages of development by Teva Pharmaceuticals Ltd. for Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with Crohn's disease for at least 3 months prior to screening.
2. Moderate to severe Crohn's disease patients as determined by the CDAI score

Exclusion Criteria:

1. Subjects who have had recent bowel surgery
2. Subjects with clinically significant GI obstructive symptoms
3. Subjects with a clinically significant or unstable medical or surgical condition
4. Subjects with unstable doses of standard of care medications (5-ASA, antibiotics, oral corticosteroids, immunosuppressants )
5. Women who are pregnant or nursing or who intend to be during the study period.
6. Women of child-bearing potential who do not practice an acceptable method of birth control

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety, Tolerability, Clinical Effect - proportion of subjects in clinical remission, proportion of subjects who respond to treatment. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Geert D'Haens, MD PhD, Principal Investigator — Imelda General Hospital
Locations (34):
- Belgium (3):
  - Teva Investigational Site 3711, Bonheiden
  - Teva Investigational Site 3712, Leuven
  - Teva Investigational Site 3713, Roeselare
- France (6):
  - Teva Investigational Site 5351, Amiens
  - Teva Investigational Site 5352, Clichy
  - Teva Investigational Site 5353, La Tronche
  - Teva Investigational Site 5350, Lille
  - Teva Investigational Site 5354, Nice
  - Teva Investigational Site 5355, Paris
- Israel (6):
  - Teva Investigational Site 8046, Jerusalem, IL
  - Teva Investigational Site 8047, Petah Tikva, IL
  - Teva Investigational Site 8050, Ramat Gan, IL
  - Teva Investigational Site 8051, Rehovot, IL
  - Teva Investigational Site 8049, Tel Aviv, IL
  - Teva Investigational Site 8048, Haifa
- Italy (3):
  - Teva Investigational Site 3069, Roma
  - Teva Investigational Site 3070, Roma
  - Teva Investigational Site 3072, San Donato Milanese (MI)
- Netherlands (2):
  - Teva Investigational Site 3819, Amsterdam
  - Teva Investigational Site 3820, Rotterdam
- Poland (4):
  - Teva Investigational Site 5361, Krakow
  - Teva Investigational Site 5360, Warsaw
  - Teva Investigational Site 5362, Wroclaw
  - Teva Investigational Site 5363, Wroclaw
- South Africa (3):
  - Teva Investigational Site 9009, Claremont, Cape Town
  - Teva Investigational Site 9017, Overport, Durban
  - Teva Investigational Site 9013, Panorama, Cape Town
- Spain (3):
  - Teva Investigational Site 3158, Barcelona
  - Teva Investigational Site 3164, Córdoba
  - Teva Investigational Site 3160, Madrid
- United Kingdom (4):
  - Teva Investigational Site 3428, Bristol
  - Teva Investigational Site 3430, Coventry
  - Teva Investigational Site 3429, Liverpool
  - Teva Investigational Site 3432, London

REFERENCES:
- [Derived] D'Haens G, Sandborn WJ, Colombel JF, Rutgeerts P, Brown K, Barkay H, Sakov A, Haviv A, Feagan BG; Laquinimod for Crohn's Disease Investigators. A phase II study of laquinimod in Crohn's disease. Gut. 2015 Aug;64(8):1227-35. doi: 10.1136/gutjnl-2014-307118. Epub 2014 Oct 3. PMID 25281416